CLINICAL TRIAL: NCT05384405
Title: Accelerated Intermittent Theta Burst Stimulation for the Treatment of Non-suicidal Self-injury in Patients With Unipolar Depression and Bipolar Depression: a Sham-controlled Study
Brief Title: aiTBS for Relieving NSSI in Depressive Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS20220425
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial testing iTBS versus sham
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active stimulation (Active Comparator): Active Intermittent theta burst stimulation to the dorsolateral prefrontal cortex; 5 sessions per day, for 5 days.
  Interventions: Device: Active iTBS
- Sham stimulation (Sham Comparator): Sham stimulation to the dorsolateral prefrontal cortex; 5 sessions per day, for 5 days.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Active iTBS — MagPro X100
  Arms: active stimulation
Device: Sham iTBS — MagPro X100
  Arms: Sham stimulation

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) has been successfully used to help patients with treatment resistant depression. However, its role in alleviating self injuries without suicidal ideation remained uncertain. This trial will compare the effectiveness of active accelerated intermittent theta burst stimulation (aiTBS) rTMS to a placebo control on non-suicidal self injury (NSSI) in patients with unipolar disorder and bipolar disorder.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of aiTBS in unipolar and bipolar depressive patients with NSSI or suicidal thoughts and behaviors by measuring changes in clinical ratings at baseline, after all the treatments, and 2 weeks, 4 weeks after treatment. 60 inpatients will be randomized to receive active or sham interventions administered to the left dorso-lateral prefrontal cortex. The treatment will apply active aiTBS rTMS involving 1800 pulses (9 minutes), 5x daily at 60 minutes intervals for 5 days. Changes in mood and sleep from baseline to the end of the study will be measured with The Hamilton Rating Scale for Depression-17 item (HAM-D17), Hamilton Anxiety Scale (HAMA), Young's Mania Scale (YMRS), and Pittsburgh Sleep Quality Index (PSQI) . Non-suicidal self injury will be assessed by the Deliberate Self-Harm Inventory (DSHI) and the Ottawa self-injury inventory (OSI). Suicidal ideation and behaviors assessments include Beck Suicidal Scale Inventory (BSI), the Ottawa self-injury inventory (OSI) and several questions from Self-Injurious Thoughts and Behaviors Interview - Revised (SITBI-R). Improvement of cognitive dysfunction could be measured by Barratt Impulsiveness Scale-11 (BIS-11), near infrared spectroscopy (fNIRS). Treatment Emergent Symptom Scale (TESS) would be used to eliminate side effects of combined drugs at baseline and the adverse event record form (AERF) will be used to appraise the safety of aiTBS treatment using these parameters. To record the change in sensitivity to pain and examine the tolerability of the treatment for these participants, visual analogue scale (VAS) is employed after completing 5 sessions treatment every day.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of DSM-5 criteria for current major depressive disorder (MDD) or bipolar disorder (BD) will be required for study entry.
2. Ages between 12 and 18 years
3. At least 1 caregivers to supervise the patient within 3 month.
4. A score of greater than 17 on the HAM-D17.
5. Occurrences of self injury behavior consistent with the DSM-5 criteria of NSSI more than 3 times in a month.
6. Willingness to participate in the study and sign informed consents

Exclusion Criteria:

1. Substance abusers such as psychoactive drugs or alcohol.
2. Severe physical disability and unable to complete follow-up.
3. Comorbid other major mental illnesses that meet the DSM-5 criteria, such as schizophrenia, mental retardation, dementia, severe cognitive impairment, attention deficit hyperactivity disorder, etc.
4. Currently in a manic episode, YMRS>12; rapid-cycling bipolar disorder, bipolar disorder with mixed features.
5. Suffering from any severe physical disease, neurological disease, traumatic brain injury, etc, that affects the structure or function of the brain in the lifetime.
6. Unable to read, understand and complete the assessment or to cooperate with the investigators.
7. Any implants covering a pacemaker, metallic or magnetic objects in the body, or other conditions not suitable for rTMS.
8. A history or family history of epilepsy and other contraindications to TMS.
9. Daily use of benzodiazepines (more than 2mg/d), theophylline, stimulants such as methylphenidate, anticonvulsants, bupropion, etc.
10. Those who have received systematic psychotherapy (interpersonal relationship therapy, dynamic therapy, cognitive behavioral therapy) within 3 months before baseline.
11. Other examination abnormalities considered to be inappropriate by investigators.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in the Deliberate Self-Harm Inventory (DSHI) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Containing one subscale ranging from 0 to 57 to measure the frequencies of NSSI behavior and one subscale ranging from 0 to 76 to measure the severity of NSSI behavior.

SECONDARY OUTCOMES:
Changes in Pittsburgh Sleep Quality Index (PSQI) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 0-21, higher score indicates severe poorer sleep quality
Changes in Hamilton Anxiety Scale (HAMA) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 0-56, higher score indicates more severe symptoms
Changes in Young's Mania Scale (YMRS) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 0-60, higher score indicates more severe symptoms
Changes in Barratt Impulsiveness Scale-11 (BIS-11) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 26-104, higher score indicates higher impulsivity
Changes in cerebral blood flow of PFC through Near Infrared Spectroscopy (fNIRS) | Baseline, after 5 treatment days
  Measuring the hemoglobin concentration of cerebral cortex during resting state and verbal fluency test.
Changes in the 17-item Hamilton Rating Scale for Depression (HAMD-17) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  This will be measured as both a continuous variable (scores on HAMD-17 ) and a categorical one (i.e. the response rates of >50% reduction from baseline HAMD-17 and remission rates defined as HAMD-17 <7).
Changes in Beck Suicidal Scale Inventory (BSI) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 0- 38, higher score indicates more severe suicide ideation.
Changes in The Clinical Global Impression (CGI) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Measuring the symptom severity, overall improvement, and therapeutic response to intervention.
Changes in the subscale of addiction of NSSI from OSI (Ottawa self-injury inventory) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 0- 28, higher score indicates higher addiction.
Changes in number of occurrences of Non-Suicidal Self Injurious ideation Through SITBI-R | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  The frequency of NSSI thoughts during the latest week
Changes in likelihood of future Non-Suicidal Self Injury Through SITBI-R | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 0-4, higher score indicates more likelihood to conduct NSSI in the future
Changes in the Deliberate Self-Harm Inventory-ideation (DSHI-ideation) | Baseline, after 5 treatment days, 2 week and 4 week post-treatment
  Range from 0 to 57 to measure the frequency of NSSI ideation

OTHER OUTCOMES:
The retrospect of NSSI behavior | Baseline
  Measured by Ottawa self-injury inventory (OSI), including reasons, addiction, site of NSSI, etc.
Borderline features of patients with NSSI | Baseline
  Measured by The Borderline Personality Feature Scale for Children - 11 (BPFS-C-11) ranging from 24 to 120
Child maltreatment of patients with NSSI | Baseline
  Measured by the Childhood Trauma Questionnaire (CTQ) ranging from 25 to 125.
Fundelmental parental style of caregivers of patients with NSSI | Baseline
  Measured by the Parental Bonding Instrument (PBI) containing two subscales ranging from 0 to 75 for both mother and father version.
Safety and tolerance of the intervention | After 5 treatment days
  Recording any side effects in the adverse event record form (AERF).

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of Second Xiangya Hospital,CSU, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No